CLINICAL TRIAL: NCT05753254
Title: Effect on Markers of Cardiovascular, Reproductive and Cancer Risk From Firefighting Activities - a Study Under Different Training Methods
Brief Title: Effect on Markers of Cardiovascular, Reproductive and Cancer Risk From Firefighting Training
Acronym: BIOBRAND3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: University of Copenhagen (Other); University Hospital Bispebjerg and Frederiksberg (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Maria Helena Guerra Andersen, Researcher, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 72403; FFIKA WP4.3 (Other Grant/Funding Number: Danish Government); AMFF 16-2022-03 (Other Grant/Funding Number: Working Environment Research Fund, Ministry of Employment); H-21068847 (Other: Danish Committee on Health Research Ethics)
Record Dates: First submitted 2023-02-02; First posted 2023-03-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Reactive Hyperemia; Micro RNA; Heart Rate Variability; DNA Strand Breaks; Oxidative Stress; Heat Stress
Keywords: Comet assay; 8-oxodG; PAH CALUX; hydroxyl-PAHs and nitro-PAH metabolites; microRNA; AhR activation; scrotal temperature; core body temperature; urine; serum; blood; follicle-stimulating hormone; inhibin B; EndoPAT
MeSH Terms: conditions — Hyperemia; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Participants will perform firefighting full day exercises under 3 different conditions (without fire, under wood fire and under gas fire), sessions which will occur with weeks in between, and biological markers will be assessed and compared in relation to a baseline session, where the participants are having theoretical classes.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind the participants to the different scenarios, neither the field staff, but all the samples will be blinded for the subsequent laboratory analysis, namely blood analysis, urine analysis, wipe samples analysis will all be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Baseline session (No Intervention): Baseline measurements will be performed in the same schedule as measurements in the three other arms. In the baseline session, participants are in classroom before starting any firefighting exercise
- Firefighting exercises without fire (Experimental): Firefighting equivalent work, with exercises performed in a clean environment, without fire (no ambient temperature, soot or smoke). This type of exercise usually precedes or complements the training under real fire conditions.
  Interventions: Other: Firefighting training exercises with no fire
- Firefighting under wood fire (Experimental): Firefighting under wood fire, with exposure to ambient heat, smoke and soot. This is the most common training scenario used in the training centres. The participants will be in teams performing pre-defined tasks (knocking down the fire, moving heavy objects, and searching and rescuing metal stand in models
  Interventions: Other: Firefighting training exercises under wood fire
- Firefighting under gas fire (Experimental): Firefighting under gas fire, with exposure to ambient heat, and expectably less smoke and soot than with wood fire. These conditions are used in some Danish training centres, with logistical advantages (ease of turning or putting out the fire and managing the fire fuel) and unknown effect relating to exposure prevention (smoke and soot). The participants will be in teams performing pre-defined tasks (knocking down the fire, moving heavy objects, and searching and rescuing metal stand in models
  Interventions: Other: Firefighting training exercises under gas fire

INTERVENTIONS:
Other: Firefighting training exercises with no fire — The participants will be performing firefighting equivalent work in a clean environment, without fire (no ambient temperature, soot or smoke).
  Arms: Firefighting exercises without fire
Other: Firefighting training exercises under wood fire — The participants will be in teams performing pre-defined tasks (knocking down the fire, moving heavy objects, and searching and rescuing metal stand in models), under wood fire conditions.
  Arms: Firefighting under wood fire
Other: Firefighting training exercises under gas fire — The participants will be in teams performing pre-defined tasks (knocking down the fire, moving heavy objects, and searching and rescuing metal stand in models), under gas fire conditions.
  Arms: Firefighting under gas fire

SUMMARY:
Epidemiological studies based on Danish registries have observed that Danish male firefighters have more cardiovascular disease, infertility diagnose and a trend to increased risk of cancer than other Danish employed males. Firefighting activities include a combination of stressors such as strenuous work under heat, smoke and soot known to be able to affect cardiovascular and reproductive health, with smoke and soot also being known to increase the risk of cancer.

The training facilities of real-fire extinguishing exercises in Denmark operate using wood or natural gas fire, which will have differential gradients of smoke, soot and possibly heat. The investigators will use different training conditions to create gradients of the different stressors and investigate health effects thereof. With this approach, the investigators expect to be able to evaluate the individual contribution of the different stressors in markers of cardiovascular, cancer and reproductive health risk. The project will include approx. 35 young conscript participants on a firefighting course, followed in four sessions, three firefighting training sessions under different fire conditions (no fire, wood fire and gas fire) and one control scenario.

DETAILED DESCRIPTION:
The study methodology is based on a crossover design on firefighting training under different conditions, with characterization of exposure and assessment of cardiovascular, cancer and reproductive effect biomarkers. The study will be performed in cooperation with the Danish Emergency Management Agency.

The study will have one baseline session, while conscripts are in a classroom, and three sessions of firefighting-related exercises under different fire conditions, used currently in firefighting training programs in Denmark. The three firefighting training sessions will be controlled for equivalent work exercise using full protective gear and under different ambient conditions of firefighting training:

* Firefighting equivalent work (no fire), with exercises performed in a clean environment, without fire (no ambient temperature, soot or smoke). This type of exercise precedes or complements the training under real fire conditions.
* Firefighting under wood fire (wood fire), with exposure to ambient heat, smoke and soot. This is the most common training scenario used by Danish Emergency Management Agency training centres.
* Firefighting under gas fire (gas fire), with exposure to ambient heat, and expectably less smoke and soot than with wood fire. These conditions are used in some Danish training centres, with logistical advantages (ease of turning or putting out the fire and managing the fire fuel) and unknown effect relating to exposure prevention (smoke and soot).

The order of the firefighting sessions will be as randomized as possible, and according to a selection of three sequence order options (no-wood-gas; wood-gas-no and gas-wood-no). Each campaign (corresponding to each rescue course) would desirably have one of these session sequences. It is not possible to blind the participants to the different scenarios, neither the field staff, but all the samples will be blinded for the subsequent laboratory analysis. The training sessions will have 1-3 weeks in between (accordingly with programmatic educational course schemes).

ELIGIBILITY:
The participants will be volunteers (both males and females) recruited among conscripts in training in a desirable involved group up to 35 individuals.

Inclusion Criteria:

* legally competent,
* conscript subjects following a Rescue Specialist Educational course

Exclusion Criteria:

* current smoking status,
* pregnancy,
* on prescribed medication,
* body mass index (BMI) bellow 19 or over 30,
* alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Change in reactive hyperemia index - afternoon | Baseline afternoon measurement, afternoon measurement immediately after firefighting without fire, afternoon measurement immediately after firefighting under wood fire and afternoon measurements immediately after firefighting under gas fire
  Reactive hyperemia index (RHI) measured with the device EndoPAT 2000. A reactive hyperemia is induced by a blood cuff on the upper arm and the peripheral vasodilation response is assessed in the small digital vessels of a fingertip with a portable device connected to a computer, with RHI determined by an algorithm from the device, with lower index values corresponding to a worsen situation.
Change in reactive hyperemia index - morning | Baseline morning measurement, morning measurement in subsequent day after firefighting without fire, morning measurement in subsequent day after firefighting under wood fire and morning measurement in subsequent day after firefighting under gas fire
  Reactive hyperemia index (RHI) measured with the device EndoPAT 2000. A reactive hyperemia is induced by a blood cuff on the upper arm and the peripheral vasodilation response is assessed in the small digital vessels of a fingertip with a portable device connected to a computer, with RHI determined by an algorithm from the device, with lower index values corresponding to a worsen situation.
Change in Heart Rate Variability pNN50 at rest - afternoon | Baseline afternoon measurement, afternoon measurement immediately after firefighting without fire, afternoon measurement immediately after firefighting under wood fire and afternoon measurements immediately after firefighting under gas fire
  Heart rate variability (HRV) measured with the device EndoPAT 2000. The HRV is calculated using the initial 5.5 complete minutes before the cuff is applied. pNN50 is the proportion of successive NN intervals differing by more than 50 milliseconds divided by the total number of N intervals (given in percentage).
Change in Heart Rate Variability pNN50 at rest - morning | Baseline morning measurement, morning measurement in subsequent day after firefighting without fire, morning measurement in subsequent day after firefighting under wood fire and morning measurement in subsequent day after firefighting under gas fire
  Heart rate variability (HRV) measured with the device EndoPAT 2000. The HRV is calculated using the initial 5.5 complete minutes before the cuff is applied. pNN50 is the proportion of successive NN intervals differing by more than 50 milliseconds divided by the total number of N intervals (given in percentage).
Change in Heart Rate Variability RMSSD at rest - afternoon | Baseline afternoon measurement, afternoon measurement immediately after firefighting without fire, afternoon measurement immediately after firefighting under wood fire and afternoon measurements immediately after firefighting under gas fire
  Heart rate variability (HRV) measured with the device EndoPAT 2000. The HRV is calculated using the initial 5.5 complete minutes before the cuff is applied. RMSSD is the square root of the mean squared differences of successive NN intervals (given in milliseconds)
Change in Heart Rate Variability RMSSD at rest - morning | Baseline morning measurement, morning measurement in subsequent day after firefighting without fire, morning measurement in subsequent day after firefighting under wood fire and morning measurement in subsequent day after firefighting under gas fire
  Heart rate variability (HRV) measured with the device EndoPAT 2000. The HRV is calculated using the initial 5.5 complete minutes before the cuff is applied. RMSSD is the square root of the mean squared differences of successive NN intervals (given in milliseconds)
Change in Heart Rate Variability ratio LF/HF at rest - afternoon | Baseline afternoon measurement, afternoon measurement immediately after firefighting without fire, afternoon measurement immediately after firefighting under wood fire and afternoon measurements immediately after firefighting under gas fire
  Heart rate variability (HRV) measured with the device EndoPAT 2000. The HRV is calculated using the initial 5.5 complete minutes before the cuff is applied. Ratio of low frequency and high frequency bands
Change in Heart Rate Variability ratio LF/HF at rest - morning | Baseline morning measurement, morning measurement in subsequent day after firefighting without fire, morning measurement in subsequent day after firefighting under wood fire and morning measurement in subsequent day after firefighting under gas fire
  Heart rate variability (HRV) measured with the device EndoPAT 2000. The HRV is calculated using the initial 5.5 complete minutes before the cuff is applied. Ratio of low frequency and high frequency bands
Changes in levels of 8-oxodG excretion in first morning urine | Baseline, before firefighting without fire, day after firefighting without fire, before firefighting under wood fire, day after firefighting under wood fire, before firefighting under gas fire, day after firefighting under gas fire
  Oxidized nucleobase 8-oxodG will be measured in urine samples by High-performance liquid chromatography (HPLC) as marker of oxidative stress, together with creatinine, for adjusting for urine concentration. Data will be reported as nanomol 8-oxodG per millimol creatinine.
Changes in levels of DNA strand breaks in peripheral blood mononuclear cells | Baseline, before firefighting without fire, day after firefighting without fire, before firefighting under wood fire, day after firefighting under wood fire, before firefighting under gas fire, day after firefighting under gas fire
  DNA strand breaks will be measured by comet assay, and reported as number of lesions per 10^6 base pairs, transformed from percentage of DNA in tail using the calibration curve from the well-establish relationship between ionizing radiation dose and yield of strand breaks in DNA.
Changes in core temperature | Baseline day, during the day of firefighting without fire, during the day of firefighting under wood fire and during the day of firefighting under gas fire.
  Core body temperature will be assessed by an ingestible pill thermometer with data recorded and reported as time series during the period in transit.
Changes in scrotal temperature | Baseline day, during the day of firefighting without fire, during the day of firefighting under wood fire and during the day of firefighting under gas fire.
  Scrotal temperature will be assessed by skin sensor placed in the scrotum of male participants and reported as scrotal skin temperature time series.
Changes in scrotal thermoregulation | Baseline day, during the day of firefighting without fire, during the day of firefighting under wood fire and during the day of firefighting under gas fire.
  Core body temperature will be assessed by an ingestible pill thermometer and scrotal temperature will be assessed by skin sensor placed in the scrotum of male participants, to assess the thermoregulation of the scrotum during firefighting exercises. Time series of core body temperature and scrotal skin temperature will be analysed for eventual thermoregulation disruption.
Changes in levels of circulating micro RNA | Baseline, before firefighting without fire, day after firefighting without fire, before firefighting under wood fire, day after firefighting under wood fire, before firefighting under gas fire, day after firefighting under gas fire
  Circulating micro RNA candidates will be measured by RNA extraction from serum samples, reverse transcribed into complementary DNA (cDNA) and analysed with quantitative polymerase chain reaction (qPCR).
Changes in urinary potency of AhR activation | Baseline, before firefighting without fire, day after firefighting without fire, before firefighting under wood fire, day after firefighting under wood fire, before firefighting under gas fire, day after firefighting under gas fire
  The aryl hydrocarbon receptor (AhR) activation will be assessed in vitro using urine samples on the PAH CALUX (Chemical Activated LUciferase gene eXpression bioassay) reporter assay. The smoke and soot exposures are complex mixtures of compounds with potential toxic effect. Routine measurements of PAHs are usually quantified for a target list of 16 common soot elements and even less chemical species for urinary metabolites, but many other compounds are present in both soot and metabolites mixtures. The toxicity of PAHs is primarily caused through the binding to AhR, and induction of AhR related genes and subsequent toxic pathways. The outcome will be measured in the form of benzo[a]pyrene equivalence.
Changes in potency of AhR activation from skin deposits | Baseline, before firefighting without fire, immediately after firefighting without fire, before firefighting under wood fire, immediately after firefighting under wood fire, before firefighting under gas fire, immediately after firefighting under gas
  The aryl hydrocarbon receptor (AhR) activation will be assessed in vitro using wipe samples on the PAH CALUX (Chemical Activated LUciferase gene eXpression bioassay) reporter assay. The smoke and soot exposures are complex mixtures of compounds with potential toxic effect. Routine measurements of PAHs are usually quantified for a target list of 16 common soot elements, but many other compounds are present in soot mixtures. The toxicity of PAHs is primarily caused through the binding to AhR, and induction of AhR related genes and subsequent toxic pathways. The outcome will be measured in the form of benzo[a]pyrene equivalence.

SECONDARY OUTCOMES:
Changes in levels of follicle-stimulating hormone in serum | Baseline, before firefighting without fire, day after firefighting without fire, before firefighting under wood fire, day after firefighting under wood fire, before firefighting under gas fire, day after firefighting under gas fire
  Follicle-stimulating hormone (FSH) will be measured in serum samples
Changes in levels of serum inhibin B | Baseline, before firefighting without fire, day after firefighting without fire, before firefighting under wood fire, day after firefighting under wood fire, before firefighting under gas fire, day after firefighting under gas fire
  Inhibin B hormone will be measured in serum samples
Changes in urinary levels of PAH metabolites excretion | Baseline, before firefighting without fire, day after firefighting without fire, before firefighting under wood fire, day after firefighting under wood fire, before firefighting under gas fire, day after firefighting under gas fire
  The internal dose of polycyclic aromatic hydrocarbons (PAHs), that would have the contribution from different exposure routes, will be assessed in first morning urine samples and measured for 7 isomer hydroxyl-PAH compounds and 5 nitro-PAH compounds, measured by high-performance liquid chromatography (HPLC)
Changes in levels of PAHs in skin wipes from the neck | Baseline, before firefighting without fire, immediately after firefighting without fire, before firefighting under wood fire, immediately after firefighting under wood fire, before firefighting under gas fire, immediately after firefighting under gas
  Skin wipes will be sampled to determine the PAH composition of deposited soot on the neck area. The wipes will be analysed for the 16 US Environmental Protection Agency priority list of PAH compounds by HPLC.
Changes in FEV1 spirometric measurements | Baseline, immediately after firefighting without fire, immediately after firefighting under wood fire and immediately after firefighting under gas fire
  Lung function will be measured by spirometry using the Spirometer device EasyOne Air. Forced Expiratory Volume at 1 second (FEV1).
Changes in FVC spirometric measurements | Baseline, immediately after firefighting without fire, immediately after firefighting under wood fire and immediately after firefighting under gas fire
  Lung function will be measured by spirometry using the Spirometer device EasyOne Air. Forced Vital capacity (FVC).
Changes in PEF spirometric measurements | Baseline, immediately after firefighting without fire, immediately after firefighting under wood fire and immediately after firefighting under gas fire
  Lung function will be measured by spirometry using the Spirometer device EasyOne Air. Peak Expiratory Flow (PEF).
Changes in FEV1/FVC ratio from spirometric measurements | Baseline, immediately after firefighting without fire, immediately after firefighting under wood fire and immediately after firefighting under gas fire
  Lung function will be measured by spirometry using the Spirometer device EasyOne Air. Forced Expiratory Volume at 1 second (FEV1) and Forced Vital Capacity (FVC) ratio is calculated from device output.
Changes in blood troponin levels | Baseline, before firefighting without fire, day after firefighting without fire, before firefighting under wood fire, day after firefighting under wood fire, before firefighting under gas fire, day after firefighting under gas fire
  Cardiac troponin levels using ELISA immunoassays will be assessed in serum samples.
Changes in work load measured by muscle activity | Baseline day, firefighting without fire day, firefighting under wood fire day and firefighting under gas fire day
  Muscle activity will be assessed to control for body workload through electromyography (EMG) using the portable device Nexus10. Bipolar surface EMG electrodes are applied to the skin over the muscles in 3 relevant body regions (shoulder, leg and back). The signals are collected with a data logger and reported as work load during a working day.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Helena G Andersen, PhD, Principal Investigator — The National Research Centre for the Working Environment (NRCWE)
Locations (2):
- Denmark (2):
  - The National Research Centre for the Working Environment, Copenhagen
  - Maria Helena Guerra Andersen, København Ø

IPD SHARING:
Plan to Share IPD: No
Supportive information and fully anonymized information will be shared and whenever possible (in supplementary material) published along with the results, but following European Union General Data Protection Regulation (GDPR) and Danish rules, no non or pseudo anonymized data might be shared.

REFERENCES:
- [Background] Andersen MHG, Saber AT, Pedersen PB, Loft S, Hansen AM, Koponen IK, Pedersen JE, Ebbehoj N, Norskov EC, Clausen PA, Garde AH, Vogel U, Moller P. Cardiovascular health effects following exposure of human volunteers during fire extinction exercises. Environ Health. 2017 Sep 6;16(1):96. doi: 10.1186/s12940-017-0303-8. PMID 28877717
- [Background] Andersen MHG, Saber AT, Clausen PA, Pedersen JE, Lohr M, Kermanizadeh A, Loft S, Ebbehoj N, Hansen AM, Pedersen PB, Koponen IK, Norskov EC, Moller P, Vogel U. Association between polycyclic aromatic hydrocarbon exposure and peripheral blood mononuclear cell DNA damage in human volunteers during fire extinction exercises. Mutagenesis. 2018 Feb 24;33(1):105-115. doi: 10.1093/mutage/gex021. PMID 29045708
- [Background] Andersen MHG, Saber AT, Pedersen JE, Pedersen PB, Clausen PA, Lohr M, Kermanizadeh A, Loft S, Ebbehoj NE, Hansen AM, Kalevi Koponen I, Norskov EC, Vogel U, Moller P. Assessment of polycyclic aromatic hydrocarbon exposure, lung function, systemic inflammation, and genotoxicity in peripheral blood mononuclear cells from firefighters before and after a work shift. Environ Mol Mutagen. 2018 Jul;59(6):539-548. doi: 10.1002/em.22193. Epub 2018 May 15. PMID 29761929
- [Background] Andersen MHG, Saber AT, Frederiksen M, Clausen PA, Sejbaek CS, Hemmingsen CH, Ebbehoj NE, Catalan J, Aimonen K, Koivisto J, Loft S, Moller P, Vogel U. Occupational exposure and markers of genetic damage, systemic inflammation and lung function: a Danish cross-sectional study among air force personnel. Sci Rep. 2021 Sep 9;11(1):17998. doi: 10.1038/s41598-021-97382-5. PMID 34504215
- [Background] Beitel SC, Flahr LM, Hoppe-Jones C, Burgess JL, Littau SR, Gulotta J, Moore P, Wallentine D, Snyder SA. Assessment of the toxicity of firefighter exposures using the PAH CALUX bioassay. Environ Int. 2020 Feb;135:105207. doi: 10.1016/j.envint.2019.105207. Epub 2019 Dec 4. PMID 31812113
- [Background] Henriksen T, Weimann A, Larsen EL, Poulsen HE. Quantification of 8-oxo-7,8-dihydro-2'-deoxyguanosine and 8-oxo-7,8-dihydro-guanosine concentrations in urine and plasma for estimating 24-h urinary output. Free Radic Biol Med. 2021 Aug 20;172:350-357. doi: 10.1016/j.freeradbiomed.2021.06.014. Epub 2021 Jun 22. PMID 34166769
- [Background] Hjollund NH, Storgaard L, Ernst E, Bonde JP, Olsen J. Impact of diurnal scrotal temperature on semen quality. Reprod Toxicol. 2002 May-Jun;16(3):215-21. doi: 10.1016/s0890-6238(02)00025-4. PMID 12128094
- [Background] Jung A, Schuppe HC. Influence of genital heat stress on semen quality in humans. Andrologia. 2007 Dec;39(6):203-15. doi: 10.1111/j.1439-0272.2007.00794.x. PMID 18076419
- [Background] Kales SN, Soteriades ES, Christophi CA, Christiani DC. Emergency duties and deaths from heart disease among firefighters in the United States. N Engl J Med. 2007 Mar 22;356(12):1207-15. doi: 10.1056/NEJMoa060357. PMID 17377158
- [Background] Keir JLA, Akhtar US, Matschke DMJ, Kirkham TL, Chan HM, Ayotte P, White PA, Blais JM. Elevated Exposures to Polycyclic Aromatic Hydrocarbons and Other Organic Mutagens in Ottawa Firefighters Participating in Emergency, On-Shift Fire Suppression. Environ Sci Technol. 2017 Nov 7;51(21):12745-12755. doi: 10.1021/acs.est.7b02850. Epub 2017 Oct 18. PMID 29043785
- [Background] Kumar K, Trzybulska D, Tsatsanis C, Giwercman A, Almstrup K. Identification of circulating small non-coding RNAs in relation to male subfertility and reproductive hormones. Mol Cell Endocrinol. 2019 Jul 15;492:110443. doi: 10.1016/j.mce.2019.05.002. Epub 2019 May 8. PMID 31077744
- [Background] Morup N, Rajpert-De Meyts E, Juul A, Daugaard G, Almstrup K. Evaluation of Circulating miRNA Biomarkers of Testicular Germ Cell Tumors during Therapy and Follow-up-A Copenhagen Experience. Cancers (Basel). 2020 Mar 23;12(3):759. doi: 10.3390/cancers12030759. PMID 32210101
- [Background] Pedersen JE, Ugelvig Petersen K, Ebbehoj NE, Bonde JP, Hansen J. Incidence of cardiovascular disease in a historical cohort of Danish firefighters. Occup Environ Med. 2018 May;75(5):337-343. doi: 10.1136/oemed-2017-104734. Epub 2018 Jan 26. PMID 29374097
- [Background] Petersen KU, Hansen J, Ebbehoej NE, Bonde JP. Infertility in a Cohort of Male Danish Firefighters: A Register-Based Study. Am J Epidemiol. 2019 Feb 1;188(2):339-346. doi: 10.1093/aje/kwy235. PMID 30452532
- [Background] Kirstine Ugelvig Petersen K, Pedersen JE, Bonde JP, Ebbehoej NE, Hansen J. Long-term follow-up for cancer incidence in a cohort of Danish firefighters. Occup Environ Med. 2018 Apr;75(4):263-269. doi: 10.1136/oemed-2017-104660. Epub 2017 Oct 21. PMID 29055884
- [Background] Pieterse B, Felzel E, Winter R, van der Burg B, Brouwer A. PAH-CALUX, an optimized bioassay for AhR-mediated hazard identification of polycyclic aromatic hydrocarbons (PAHs) as individual compounds and in complex mixtures. Environ Sci Technol. 2013 Oct 15;47(20):11651-9. doi: 10.1021/es403810w. Epub 2013 Sep 25. PMID 23987121
- [Background] Schwartz C, Bolling AK, Carlsten C. Controlled human exposures to wood smoke: a synthesis of the evidence. Part Fibre Toxicol. 2020 Oct 2;17(1):49. doi: 10.1186/s12989-020-00375-x. PMID 33008417
- [Background] Alhamdow A, Lindh C, Albin M, Gustavsson P, Tinnerberg H, Broberg K. Early markers of cardiovascular disease are associated with occupational exposure to polycyclic aromatic hydrocarbons. Sci Rep. 2017 Aug 25;7(1):9426. doi: 10.1038/s41598-017-09956-x. PMID 28842704